CLINICAL TRIAL: NCT03130985
Title: PREventive Left Atrial appenDage Resection for predICtion of fuTure Atrial Fibrillation
Brief Title: Tissue, Blood and Biomarkers to Predict Future Atrial Fibrillation
Acronym: PREDICT-AF
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, J.R. de Groot, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL50754.018.14
Record Dates: First submitted 2015-06-04; First posted 2017-04-27 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Atrial Fibrillation
Keywords: microRNA; biomarker
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Left atrial appendages will be deep frozen and fixed Plasma samples and whole blood will be collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac surgery patients: The study cohort will comprise of patients without a history of AF that undergo cardiac surgery (CABG or mitral valve surgery) with increased CHADSVASC scores of ≥2.

SUMMARY:
Patients undergoing coronary artery bypass grafting (CABG), aortic (valve) or mitral valve surgery are at risk of developing postoperative and new-onset atrial fibrillation (AF), but adequate risk prediction is currently impossible. This study aims to discover tissue and circulating microRNAs and protein biomarkers that may help to unravel the pathophysiological processes underlying AF and are potential tools for risk stratification and prognosis or may become future targets of therapy.

This study will be a single-center cohort study of 150 patients undergoing cardiac surgery, which will constitute the beginning of the follow-up period. Left atrial appendages, whole blood and epicardial mappings will be collected. Patients will be followed for 2 years with regular holter investigations to detect postoperative and new-onset AF.

DETAILED DESCRIPTION:
Study procedures:

The left atrial appendage (LAA) will be removed for research and intended prophylactic purposes, using a surgical stapler or surgical knife prior to the standard procedure. Epicardial mappings may be performed during cardiac surgery with a 48-multi-electrode. Patients will be followed with regular 24-hour Holter investigations.

This study will be an exploratory study with a required inclusion of 150 patients, based on the estimated event rate. Patients will be recruited by the investigators during pre-operative assessment.

Clinical data will be gathered at baseline and stored in a customized microsoft access entry database. Statistical analysis will be performed in collaboration with the Bioinformatics Laboratory from the Academic Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Elective sternotomy for either coronary artery bypass surgery or aortic (valve) surgery or mitral valve surgery
* CHA2DS2 VASC score ≥ 2
* Sinus rhythm
* Age between 18 and 80 years
* Legally competent and willing and able to sign informed consent

Exclusion Criteria:

* Unable or unwilling to comply with study procedures
* Documented or reported history of atrial fibrillation, atrial flutter (duration > 5 minutes) or ventricular tachycardia
* Emergency or redo of CABG
* Emergency valvular surgery or pericarditis or endocarditis
* NYHA class IV heart failure symptoms or left ventricular ejection fraction < 35%
* Pregnancy or of childbearing potential without adequate contraception
* History of previous radiation therapy of the thorax
* Active malignancy
* Active inflammtion or auto-immune disease
* Surgery for congenital anomalies
* Circumstances that prevent follow-up (no permanent home or address, transient, etc.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients are eligible that are referred to the investigators' tertiary cardiothoracic center for mitral valve surgery, (aortic) valve surgery or coronary artery bypass surgery and meet in- and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-05-12 (Actual); Primary Completion 2020-07-06 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
incident Atrial Fibrillation | within 2 years after surgery
  A de novo 30 second continuous rhythm registration of AF, or an ECG recording of an AF episode within 2 years after surgery (with a blanking period for the postoperative period <30 days).
Postoperative Atrial Fibrillation | within the first 30 days after surgery
  A 30 second continuous rhythm registration of AF, or an ECG recording of an AF episode in the first 30 days following cardiac surgery or registered at the first 24h Holter monitoring if scheduled within 6 weeks following cardiac surgery.

SECONDARY OUTCOMES:
Quality of Life defined by 36-Item Short Form Health Survey questionnaire | at 6 months and 1 year follow-up
  The quality of life is measured by 36-Item Short Form Health Survey questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Joris de Groot, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] van den Berg NWE, Neefs J, Kawasaki M, Nariswari FA, Wesselink R, Fabrizi B, Jongejan A, Klaver MN, Havenaar H, Hulsman EL, Wintgens LIS, Baalman SWE, Meulendijks ER, van Boven WJ, de Jong JSSG, van Putte BP, Driessen AHG, Boersma LVA, de Groot JR; PREDICT-AF Investigators. Extracellular matrix remodeling precedes atrial fibrillation: Results of the PREDICT-AF trial. Heart Rhythm. 2021 Dec;18(12):2115-2125. doi: 10.1016/j.hrthm.2021.07.059. Epub 2021 Jul 29. PMID 34332113
- [Derived] van den Berg NWE, Neefs J, Berger WR, Boersma LVA, van Boven WJ, van Putte BP, Kaya A, Kawasaki M, Driessen AHG, de Groot JR; PREDICT AF Investigators. PREventive left atrial appenDage resection for the predICtion of fuTure atrial fibrillation: design of the PREDICT AF study. J Cardiovasc Med (Hagerstown). 2019 Nov;20(11):752-761. doi: 10.2459/JCM.0000000000000868. PMID 31567634